CLINICAL TRIAL: NCT02523989
Title: The Relationship Between Genetic Polymorphism of Arsenic Methylation Enzymes, Arsenic Methylation Capability and Blood Metals, and Developmental Delays in Preschool Children
Brief Title: The Relationship Between Arsenic Methylation Capability and Blood Metals in Children With Developmental Delays
Status: Completed | Type: Observational
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Associate Professor, Taipei Medical University
Other Study IDs: SKH-TMU-100-06
Record Dates: First submitted 2015-08-07; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Developmental Delays
Keywords: arsenic; heavy metal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Blood and urine samples of participants were collected and urine used for the analysis of the arsenic species using high performance liquid chromatography linked hydride generator and atomic absorption spectrometry. Buffy coat were separated from plasma and extract DNA to analyze the genetic polymorphism of arsenic methylation related enzymes using polymerase chain reaction and restriction fragment length polymorphism. 2 ml blood were digested for the determination of mercury, lead and arsenic.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- study group: children confirmed to have developmental delays
  Interventions: Other: study group
- control group: children with typical development
  Interventions: Other: study group

INTERVENTIONS:
Other: study group — Explore the relationship of heavy metals and health related quality of life, including the relationship between the developmental delays and polymorphism of arsenic methylation enzymes, arsenic methylation capability and blood metals. Identify the interaction of children function, health condition, and quality of life and arsenic methylation and blood metals in children with developmental delays.

SUMMARY:
The purpose of this study is to explore the relationship between arsenic methylation and blood metals in children with developmental delays and its correlation with health related quality of life.

DETAILED DESCRIPTION:
The investigators recruited children with developmental delays and children with normal development from Shin-Kong Ho-Su Memorial Hospital as controls. Information obtained from the interview included socioeconomic and basic demographic characteristics as well as children function, health condition, and quality of life. On the other hand, blood and urine samples of the participants were collected for the analysis of arsenic methylation related enzymes using polymerase chain reaction and restriction fragment length polymorphism. 2 ml blood were digested for the determination of mercury, lead and arsenic. The relationship between arsenic methylation and blood metals in children with developmental delays and its correlation with health related quality of were analyzed.

ELIGIBILITY:
Study group:

Inclusion Criteria:

* children with developmental delays obtained written informed consent from parents

Exclusion Criteria:

* parents refused for participation of their children to the intervention failed to obtain the written informed consent from parents

Control group:

Inclusion Criteria:

* children with normal development obtained written informed consent from parents

Exclusion Criteria:

* parents refused for participation of their children to the intervention failed to obtain the written informed consent from parents

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children with developmental delays and children with normal development
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
heavy metal assessment | 3 months
  laboratory analysis

SECONDARY OUTCOMES:
quality of life | 2 weeks
  questionnaires analysis

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Visiting staff
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan